CLINICAL TRIAL: NCT02137538
Title: Randomization to Letrozole vs. Anastrozole in Short Pubertal Males
Brief Title: Aromatase Inhibitor Growth Study: Letrozole vs. Anastrozole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Laura K Bachrach, Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI growth study
Record Dates: First submitted 2014-05-05; First posted 2014-05-14 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Short Stature
MeSH Terms: conditions — Dwarfism | interventions — Letrozole; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letrozole (Active Comparator): Letrozole 2.5 mg daily
  Interventions: Drug: Letrozole
- Anastrozole (Active Comparator): Anastrozole 1 mg daily
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Letrozole
  Arms: Letrozole
Drug: Anastrozole
  Arms: Anastrozole

SUMMARY:
The purpose of the study is to determine if there are differences in the final height or hormone profile of short pubertal boys placed on different forms of aromatase inhibitor now routinely used to increase stature: Anastrozole and Letrozole. It also should determine if there are differences in the side effect profiles of the two drugs to be used.

ELIGIBILITY:
Inclusion Criteria:

* Current height less than 5th percentile AND/OR
* Predicted adult height (based on bone age) more than 10 cm below target height (mid parental height)
* Evidence of puberty: physical signs and serum luteinizing hormone > 0.3 IU/L and testosterone > 15 ng/dl

Exclusion Criteria:

* Bone age reading more than 14.0 years
* Follicle stimulating hormone > 20 IU/L

Ages: 10 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2009-11-18 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E Kirk Neely, MD, Principal Investigator — Stanford University; Laura K Bachrach, MD, Principal Investigator — Stanford University; Walter A Zegarra, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neely EK, Kumar RB, Payne SL, Ranadive SA, Suchet DI. Letrozole vs anastrozole for height augmentation in short pubertal males: first year data. J Clin Endocrinol Metab. 2014 Nov;99(11):4086-93. doi: 10.1210/jc.2014-2432. Epub 2014 Aug 19. PMID 25137428

RESULTS

PARTICIPANT FLOW:
Groups:
- Letrozole: Participants receive letrozole 2.5 mg daily
- Anastrozole: Participants receive anastrozole 1 mg daily
Period: Overall Study
Arm/Group | Letrozole | Anastrozole
Started | 39 | 40
Completed | 23 | 26
Not Completed | 16 | 14

BASELINE CHARACTERISTICS:
Population: Participants who finished the first year of therapy are included in the analysis, excluding participants who had received growth hormone.
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Anastrozole | Total
Number analyzed (Participants) | 30 | 35 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (1.2) | 13.9 (1.5) | 13.9 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 35 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 35 | 65
Bone age [Mean (Standard Deviation); unit: months] | 156.1 (6.6) | 156.3 (12.2) | 156.2 (9.9)
Predicted Adult Height [Mean (Standard Deviation); unit: cm] | 167.2 (5.8) | 167.3 (6.9) | 167.2 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Predicted Adult Height at Year 3
Description: Heights will be obtained by physical exam every 6 months during treatment. Skeletal maturation will be assessed from an x-ray by the method of Greulich and Pyle at baseline and every 12 months until the end of treatment.
  Predicted adult height will be calculated at baseline and at the end of treatment based upon measured height and skeletal maturation (bone age).
Time Frame: Year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
cm | 167.8 (5.8) | 169.4 (5.1)

2. Secondary Outcome: Serum Testosterone
Time Frame: Baseline, year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
ng/dL
  Baseline | 213.1 (133.7) | 162.1 (124.6)
  Year 3 | 882.3 (250.5) | 680.1 (179.5)

3. Secondary Outcome: Dihydrotestosterone
Time Frame: Baseline, year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
ng/dL
  Baseline | 22.5 (11.3) | 19.1 (9.7)
  Year 3 | 65.0 (20.2) | 44.1 (23.5)

4. Secondary Outcome: Androstenedione
Time Frame: Baseline, year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
ng/dL
  Baseline | 35.3 (13.1) | 37.4 (21.4)
  Year 3 | 79.9 (21.5) | 77.9 (28.2)

5. Secondary Outcome: Luteinizing Hormone
Time Frame: Baseline, year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
mIU/mL
  Baseline | 2.3 (1.5) | 1.8 (1.1)
  Year 3 | 4.7 (1.9) | 3.4 (2.0)

6. Secondary Outcome: Follicle Stimulating Hormone
Time Frame: Baseline, year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
mIU/mL
  Baseline | 3.3 (1.9) | 2.5 (1.3)
  Year 3 | 6.6 (2.4) | 4.5 (2.9)

7. Secondary Outcome: Insulin-like Growth Factor Type 1
Time Frame: Baseline, year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
ng/mL
  Baseline | 306.2 (112.8) | 306.9 (112.9)
  Year 3 | 226.1 (54.4) | 298.7 (78.8)

8. Secondary Outcome: Inhibin B
Time Frame: Baseline, year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
pg/mL
  Baseline | 203.4 (55.0) | 217.0 (65.2)
  Year 3 | 257.6 (61.1) | 262.1 (97.9)

9. Secondary Outcome: Estradiol
Time Frame: Baseline, year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
pg/mL
  Baseline | 4.9 (3.6) | 4.7 (4.7)
  Year 3 | 2.7 (2.1) | 6.2 (2.5)

10. Secondary Outcome: Estrone
Time Frame: Baseline, year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
pg/mL
  Baseline | 8.7 (4.8) | 8.0 (4.9)
  Year 3 | 2.7 (0.3) | 3.5 (3.2)

11. Secondary Outcome: Number of Adverse Events Related to Acne or Bone Fracture
Time Frame: 3 years
Population: as for baseline characteristics
Measure: Number; unit: events
Arm/Group | Letrozole | Anastrozole
Number analyzed (Participants) | 30 | 35
events
  Acne | 3 | 3
  Fracture | 3 | 5

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Letrozole | Anastrozole
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 2/40
Other Adverse Events (participants affected / at risk) | 12/39 | 10/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole (N=39) | Anastrozole (N=40)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unexpected serious adverse event; significant but not persistent.
Neuro event (Nervous system disorders) | 0 (0) | 1 (1) — Unexpected serious adverse event; significant but not persistent.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole (N=39) | Anastrozole (N=40)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (5)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Aggression (Nervous system disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Hair loss (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT02137538/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT02137538/SAP_001.pdf